CLINICAL TRIAL: NCT03292276
Title: Improving Hand Motor Function After Stroke: Role of Robotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, MD PhD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44/2016
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2017-09

CONDITIONS: It is Possible That Amadeo Will Guarantee a Greater Clinical Improvement as Compared to an Occupational Therapy Thanks to the Strengthening of Brain Plasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amadeo training (Experimental): All participants will receive 40 sessions of treatment (45-minute) for 8 consecutive weeks (5 days/week). The robotic exercises will be carried in passive modality (15 minutes), passive/plus (15 minutes), assisted modality (15 minutes).
  Interventions: Device: Amadeo Training
- occupational therapy (Active Comparator): All participants will receive 40 sessions of treatment (45-minute) for 8 consecutive weeks (5 days/week). The control group will receive the same amount of training by physiotherapist skilled in occupational tharapy.
  Interventions: Device: Amadeo Training

INTERVENTIONS:
Device: Amadeo Training — To understand the cortical modifications related to movement preparation and execution after robot-assisted training we will study the EEG modifications of cortical activity using time-frequency event-related EEG and task-related coherence (TRCoh).
  Friedman ANOVA with post-hoc t-test (corrected for multiple comparisons) will be used to assess the significance of training-induced changes in the two groups.

SUMMARY:
Two recent randomized clinical trials reported a significant contribute of Amadeo toward the recovery of hand motor function in acute stroke patients in association with physiotherapy and/or occupational therapy. However, no data are available in patients with chronic stroke, and the neurophysiological mechanisms underlying such clinical improvement need to be elucidated. Given that robotic devices harness brain plasticity to foster motor function recovery, a deeper understanding of the neurophysiological bases of Amadeo training could help clinician to realize patient-tailored rehabilitative training based brain plasticity knowledge. We planned a pilot randomized-controlled observer trial aimed at evaluating the effects of intensive robot-assisted hand therapy compared with intensive occupational therapy in chronic phase after stroke. We estimated that 40 patients per group will be required to demonstrate a greater effect of Amadeo as compared to occupational therapy, with an effect size of 0.5. Twenty chronic stroke patients (at their first-ever stroke) will be enrolled and randomized into two groups. The experimental group will be provided with Amadeo training. The Control group will be provided with occupational therapy executed by a trained physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke patients at their first-ever supratentorial stroke

Exclusion Criteria:

* presence of severe medical, psychiatric and cognitive abnormalities as to interfere with the treatment.
* controindications to the device use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Nine hole peg test | by 5 minutes
  Administered by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. The board should be placed at the client's midline, with the container holding the pegs oriented towards the hand being tested. Only the hand being evaluated should perform the test. Hand not being evaluated is permitted to hold the edge of the board in order to provide stability. Scores are based on the time taken to complete the test activity, recorded in seconds. Alternative scoring - the number of pegs placed in 50 or 100 seconds can be recorded. In this case, results are expressed as the number of pegs placed per second. Stopwatch should be started from the moment the participant touches the first peg until the moment the last peg hits the container.

SECONDARY OUTCOMES:
cortical modifications related to movement preparation and execution after robot-assisted training | about 30 minutes
  Assessment of EEG modifications of cortical activity using time-frequency event-related EEG and task-related coherence (TRCoh).

CONTACTS AND LOCATIONS:
Overall Officials: Placido Bramanti, Study Chair — IRCCS Neurolesi
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: No